CLINICAL TRIAL: NCT03579953
Title: Theta-Burst Stimulation As A Tool To Change Smoking Behavior
Brief Title: Nicotine TMS EFT Smoking Pilot Study
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 74722
Record Dates: First submitted 2018-06-12; First posted 2018-07-09 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Smoking; Nicotine Dependence; Addiction; Smoking, Cigarette
Keywords: Brain Stimulation
MeSH Terms: conditions — Smoking; Tobacco Use Disorder; Behavior, Addictive; Cigarette Smoking

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Real cTBS to MPFC (Experimental): One session of real cTBS treatment delivered to the medial prefrontal cortex (MPFC) (2 trains of stimulation over the MPFC as defined by EEG coordinates (FP1); each train: 120 sec, 3 pulse bursts presented at 5Hz, 15 pulses/sec, 1800 pulses/train, 60 sec intertrain interval; 110% RMT, MagPro X100 Cool Coil; 3600 pulses total).
  Interventions: Device: Real cTBS
- Sham cTBS to MPFC (Sham Comparator): One session of sham cTBS treatment delivered to the medial prefrontal cortex (MPFC) (2 trains of stimulation over the MPFC as defined by EEG coordinates (FP1); each train: 120 sec, 3 pulse bursts presented at 5Hz, 15 pulses/sec, 1800 pulses/train, 60 sec intertrain interval; 110% RMT, MagPro X100 Cool Coil; 3600 pulses total).
  Interventions: Device: Sham cTBS

INTERVENTIONS:
Device: Real cTBS — This will be delivered with the Magventure Magpro system; 3600 pulses with the active sham coil (double blinded using the USB key).
  Arms: Real cTBS to MPFC
Device: Sham cTBS — This will be delivered with the sham Magventure Magpro system; 3600 pulses with the active sham coil (double blinded using the USB key). The MagVenture MagPro system has an integrated active sham that passes current through two surface electrodes placed on the skin beneath the B60 coil.
  Arms: Sham cTBS to MPFC

SUMMARY:
Prior and recent evidence suggests a role of medial prefrontal cortex (MPFC) in cigarette smoking. Episodic Future Thinking (EFT) has also been shown to be associated with increased delayed discounting and reduced cigarette self administration. In the present study, we will examine whether a single administration of theta-burst transcranial magnetic stimulation (tbTMS) can increase Episodic Future Thinking and delayed discounting while reducing craving for nicotine.

DETAILED DESCRIPTION:
The purpose of this study is to develop theta burst transcranial magnetic stimulation (tbTMS) as a potential treatment for nicotine addiction. Theta burst TMS is a non-invasive technique that uses magnetic pulses to temporarily stimulate specific brain areas in awake people (without the need for surgery, anesthetic, or other invasive procedures). This study will test whether tbTMS over the forehead can produce a reduction in things that may prompt individuals to want to smoke cigarettes. TMS has been approved by the Food and Drug Administration as an investigational tool as well as a therapy for depression. However, TMS is not approved by the Food and Drug Administration as a treatment for nicotine cravings and other addictions.

This study consists of one consent session and one TMS session. Participants will be asked to complete a series of questionnaires and computer assessments about nicotine both before and after a single tbTMS session.

ELIGIBILITY:
Inclusion Criteria:

1. 18-65 years of age
2. Smoke at least 10 cigarettes a day (on average)
3. Not be pregnant
4. Meet all criteria on a standardized TMS safety screen (including to but not limited to implanted electronic devices, bullets or metallic fragments above the neck, hair clips that cannot be removed)
5. No barriers to making contact between the TMS coil and the skin (e.g. cornrows that cannot be removed, glasses that the participant is unwilling to remove)

Exclusion Criteria:

1. Report comorbid mental or physical illness (managed or unmanaged)
2. Currently using prescription medication that might affect smoking or nicotine metabolism
3. Using smokeless tobacco or alternative nicotine products
4. History of epilepsy or seizures (other than childhood febrile seizures)
5. History of chronic migraines

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-05-22 (Actual); Primary Completion 2019-06-10 (Actual); Study Completion 2019-06-10 (Actual)

PRIMARY OUTCOMES:
Changes in craving after a single session of cTBS | For the duration of the study, approximately 24 hours following real or sham cTBS
  The effect of real versus sham cTBS on nicotine craving will be assessed by comparing pre-TMS and post-TMS changes in nicotine craving scores.

SECONDARY OUTCOMES:
Changes in delayed discounting after a single session of cTBS | For the duration of the study, approximately 24 hours following real or sham cTBS
  The effect of real versus sham cTBS on nicotine craving will be assessed by comparing pre-TMS and post-TMS changes in delayed discounting scores.

CONTACTS AND LOCATIONS:
Overall Officials: Colleen A Hanlon, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No